CLINICAL TRIAL: NCT05022017
Title: EOS MODIC : Inflammatory Disc Disease: Description of Statics by EOS Imaging and Evaluation of the Efficacy of Intradiscal Corticosteroid Infiltration
Brief Title: Description of Statics by EOS Imaging and Evaluation of the Efficacy of Intradiscal Corticosteroid Infiltration
Acronym: EOSMODIC
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: EOS MODIC
Record Dates: First submitted 2021-04-30; First posted 2021-08-26 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Inflammatory Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inflammatory disc disease or Modic 1 disc disease is a radiological entity first described by Modic in 1988 and corresponds to an inflammatory signal on MRI defined by the presence of a T2-weighted hypersignal and a T1-weighted hyposignal of the vertebral endplates adjacent to a pathological disc.

The presence of these radiological abnormalities are significantly associated with chronic low back pain, the therapeutic management of which may include lumbar rehabilitation, rigid corset, spinal infiltrations and surgical treatment. Corticosteroid infiltration of the pathological intervertebral disc (intradiscal infiltration) has been evaluated in low back pain due to Modic 1 disc disease with short-term efficacy. The clinical response to this infiltration is not always optimal and to date in the literature, no predictive factor of response has been identified.

DETAILED DESCRIPTION:
There are several hypotheses to explain this phenomenon: mechanical, genetic, infectious or inflammatory. One of the mechanical hypotheses would be the presence of an instability of the spinal segment (hypermobility of the spinal segment) and disorders of the sagittal statics of the spine with angles of thoracic kyphosis and lumbar lordosis weak and a weak sacral slope supporting a hyperpressure passing by the discs and the genesis of discopathy.

In this work, the investigators will evaluate the different parameters of the spinal statics in the sagittal plane and in the frontal plane (sacral slope, pelvic version, Roussouly classification, cobb angle...) by EOS imaging as well as the parameters of the Modic 1 anomaly on lumbar MRI (spinal stage, Pfirmann classification, laterality of the inflammatory signal) in a population of patients who received intradiscal corticosteroid infiltration for low back pain in the context of Modic 1 disc disease.

The analysis of the different radiological parameters could enrich the investigator's understanding of the pathophysiology and evaluate radiological factors predictive of the effectiveness of intradiscal infiltration in this population. This could allow us to adapt the management of low back pain patients with Modic 1 disc disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* French speaking patient
* Patient hospitalized in the rheumatology department of GHPSJ between 01/01/2014 and 31/12/2020 for MODIC 1
* Patients who received as part of their management an intra-disc infiltration with hydrocortancyl.

Exclusion Criteria:

* Patient under guardianship or curators
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his data for this research
* Patient having benefited from another infiltration between the intradiscal infiltration and the collection of efficacy data at 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in the rheumatology department of GHPSJ between 01/01/2014 and 31/12/2020 for MODIC 1
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of the intra-disc infiltration at 3 months on the pain felt by the patient. | 3 months
  Percentage of patients with improved low back pain defined as a decrease in Visual Analogue Scale (VAS) pain >3 at 3 months after intradiscal infiltration compared to VAS at admission.
  VAS scale : minimum score 0 (no pain) / higher score 10 (greater pain intensity)

SECONDARY OUTCOMES:
Change in analgesic consumption (Level 1, Level 2, Level 3 and NSAIDs) at 3 months. | 3 months
  Consumption of level 1, 2 or 3 painkillers and NSAIDs in the previous week (number of doses per day and per week).
Describe the parameters of spinal statics in the frontal planes in Modic 1 disc disease. | 3 months
  Distribution of the values of the parameters of the spinal statics in the sagittal plane (sacral slope, pelvic incidence, pelvic version, lumbar lordosis, Roussouly classification) and in the frontal plane (cobb angle).
Compare the parameters of spinal statics according to the different stages of Modic 1 disc disease | 3 months
  Distribution of the values of spinal statics parameters in the sagittal plane (sacral slope, pelvic incidence, pelvic version, lumbar lordosis, Roussouly classification) and in the frontal plane (cobb angle) according to the presence of low lumbar (L4L5 L5S1) or high lumbar (L1L2 L2L3 L3L4) disc disease.
Predictive factors (clinical and radiological) of the effectiveness of intra-disc infiltration | 3 months
  Correlation between pain improvement 3 months after infiltration and the type of disc disease (cobb scoliosis > 10°) as well as the parameters of spinal statics in the sagittal and frontal planes and the type of disc damage according to the Pfirmann classification

CONTACTS AND LOCATIONS:
Overall Officials: Thomas HUET, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France